CLINICAL TRIAL: NCT01094782
Title: Evaluating the Effect of Acupuncture on Pain Relief Using QST
Brief Title: Evaluating the Effect of Acupuncture on Pain Relief Using Quantitative Sensory Testing (QST)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jianren Mao, MD, PhD, Director, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2009P 0001551; R01AT005819 (NIH)
Record Dates: First submitted 2010-03-19; First posted 2010-03-29 (Estimated); Results first posted 2018-07-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Pain
Keywords: Pain; Pain management
MeSH Terms: conditions — Pain; Agnosia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Healthy - True Acupuncture (Active Comparator): Healthy volunteers with no neck or back pain who attended 7 visits over 4 weeks and received 6 30 minute acupuncture treatment sessions during visits 2-7.This group received true acupuncture treatment (the needles punctured the skin).
  Interventions: Other: Acupuncture
- Healthy - Sham Acupuncture (Sham Comparator): Healthy with no neck or back pain who attended 7 visits over 4 weeks and received 6 30 minute acupuncture treatment sessions during visits 2-7. This group received sham acupuncture treatment (the needles did not puncture the skin).
  Interventions: Other: Sham Acupuncture
- Healthy - No Treatment (No Intervention): Healthy volunteers with no neck or back pain who attended 3 visits over 4 weeks and received no sham or true acupuncture treatment.
- Pain - True Acupuncture (Active Comparator): Volunteers with radiating neck or back pain who attended 7 visits over 4 weeks and received 6 30 minute acupuncture treatment sessions during visits 2-7. This group received true acupuncture treatment (the needles punctured the skin).
  Interventions: Other: Acupuncture
- Pain - Sham Acupuncture (Sham Comparator): Volunteers with radiating neck or back pain who attended 7 visits over 4 weeks and received 6 30 minute acupuncture treatment sessions during visits 2-7. This group received sham acupuncture treatment (the needles did not puncture the skin).
  Interventions: Other: Sham Acupuncture
- Pain - No Treatment (No Intervention): Volunteers with radiating neck or back pain who attended 3 visits over 4 weeks and received no sham or true acupuncture treatment.

INTERVENTIONS:
Other: Acupuncture — Subjects receive 6 acupuncture treatments for neck or back pain.
  Arms: Healthy - True Acupuncture; Pain - True Acupuncture
Other: Sham Acupuncture — Subjects receive 6 sham acupuncture treatments for neck or back pain.
  Arms: Healthy - Sham Acupuncture; Pain - Sham Acupuncture

SUMMARY:
The purpose of this study is to explore a new approach in assessing the effectiveness of acupuncture therapy in the treatment chronic pain conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Subject will be between ages 18 to 65 years. Both male and female subjects will be recruited.
2. Subject should have had cervical or lumbar radicular pain for at least two months. This requirement is to avoid the uncertainty of an unstable pain condition and to minimize the study variation.
3. Subject has a pain score of 4 or above (Visual Analog Scale (VAS): 0 - 10 from no pain to worst pain).
4. Cervical or lumbar radicular pain will include, but is not limited to, such clinical conditions as disk herniation, spinal stenosis, and post-laminectomy syndrome.
5. For controls, healthy subjects without radicular pain for at least three months will be recruited. *We are no longer accepting healthy volunteers.*

Exclusion Criteria:

1. Subject has detectable sensory deficits at the site of QST. Sensory deficits refer to such conditions resulting from neurological diseases or medical conditions causing peripheral polyneuropathy and sensory changes, which include but are not limited to diabetic neuropathy, alcoholic neuropathy, AIDS neuropathy, severe thyroid disease, and severe liver or kidney disorders.
2. Subject has scar tissue, infection, or acute injury at the site of QST.
3. Subject is on anticoagulation therapy.
4. Subject is pregnant.
5. Subject is tested positive on illicit drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Center for Translational Pain Research, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 254 participants were enrolled in the study and were randomly assigned to one of the 6 study arms at "Visit 1". 6 participants were later found to be ineligible to continue to participate (e.g. drug screen, medical history, no longer interested) further in "Visit 1" and they did not recieve study intervention.
Groups:
- Healthy - True Acupuncture: Healthy volunteers with no neck or back pain who attended 7 visits over 4 weeks and received 6 30 minute acupuncture treatment sessions during visits 2-7.
  This group received true acupuncture treatment (the needles punctured the skin).
Period: Overall Study
Arm/Group | Healthy - True Acupuncture | Healthy - Sham Acupuncture | Healthy - No Treatment | Pain - True Acupuncture | Pain - Sham Acupuncture | Pain - No Treatment
Started | 39 | 39 | 34 | 56 | 42 | 38
Completed | 31 | 29 | 31 | 45 | 31 | 30
Not Completed | 8 | 10 | 3 | 11 | 11 | 8
Not completed — Withdrawal by Subject | 5 | 5 | 1 | 5 | 5 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2 | 1 | 4
Not completed — Positive Drug Screen | 2 | 2 | 1 | 1 | 3 | 2
Not completed — Sensory Deficit at Site of QST | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Unable to Complete Questionnaires | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Healthy Subject Had Pain | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Hypertension | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Wrong Pain Condition | 0 | 0 | 0 | 2 | 1 | 1
Not completed — Recent Interventional Injection | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Low Visual Analog Scale (VAS) Score | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Noncompliance With Study Schedule | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy - True Acupuncture | Healthy - Sham Acupuncture | Healthy - No Treatment | Pain - True Acupuncture | Pain - Sham Acupuncture | Pain - No Treatment | Total
Number analyzed (Participants) | 39 | 39 | 34 | 56 | 42 | 38 | 248
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 39 | 34 | 55 | 42 | 38 | 247
  >=65 years | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 14 | 23 | 31 | 24 | 133
  Male | 19 | 18 | 20 | 33 | 11 | 14 | 115
Region of Enrollment [Number; unit: participants]
  United States | 39 | 39 | 34 | 56 | 42 | 38 | 248

OUTCOME MEASURES:

1. Primary Outcome: Heat Pain Tolerance - Baseline: Maximum Temperature (Heat) That Could be Tolerated by Participants
Description: Changes in response to heat stimulation stated as tolerance to heat. Responses are measured with a quantitative sensory testing (QST) device. Measurements were taken before the course of a 4 week acupuncture treatment schedule.
Time Frame: Start of Week 1
Population: Primary analysis was performed using the mITT (Modified Intent to Treat) method. Participants who were assigned a group and received their 1st study intervention were included in the analysis.
Measure: Mean (Standard Deviation); unit: Degrees Celcius
Arm/Group | Healthy - True Acupuncture | Healthy - Sham Acupuncture | Healthy - No Treatment | Pain - True Acupuncture | Pain - Sham Acupuncture | Pain - No Treatment
Number analyzed (Participants) | 34 | 30 | 31 | 46 | 33 | 30
Degrees Celcius | 49.9 (1.7) | 50.5 (1.3) | 49.9 (1.7) | 49.5 (2.4) | 49.7 (2.2) | 50.1 (2)

2. Primary Outcome: Heat Pain Tolerance - Visit 2 or 4: Maximum Temperature (Heat) That Could be Tolerated by Participants
Description: Changes in response to heat stimulation stated as tolerance to heat. Responses are measured with a quantitative sensory testing (QST) device. Measurements were taken during the course of a 4 week acupuncture treatment schedule. Those in the no treatment groups were attending their 2nd visit, which occured on the same timeline as if they were attending the 4th visit as a treatment group subject.
Time Frame: End of Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees Celcius
Arm/Group | Healthy - True Acupuncture | Healthy - Sham Acupuncture | Healthy - No Treatment | Pain - True Acupuncture | Pain - Sham Acupuncture | Pain - No Treatment
Number analyzed (Participants) | 34 | 30 | 31 | 46 | 33 | 30
Degrees Celcius | 49.8 (1.6) | 50.3 (1.6) | 50.2 (1.6) | 49.6 (2.8) | 50.3 (2.1) | 50.0 (2.1)

3. Primary Outcome: Heat Pain Tolerance - Visit 3 or 7: Maximum Temperature (Heat) That Could be Tolerated by Participants
Description: Changes in response to heat stimulation stated as tolerance to heat. Responses are measured with a quantitative sensory testing (QST) device. Measurements were taken after the course of a 4 week acupuncture treatment schedule. Those in the no treatment groups were attending their 3rd visit, which occured on the same timeline as if they were attending the 7th visit as a treatment group subject.
Time Frame: End of Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees Celcius
Arm/Group | Healthy - True Acupuncture | Healthy - Sham Acupuncture | Healthy - No Treatment | Pain - True Acupuncture | Pain - Sham Acupuncture | Pain - No Treatment
Number analyzed (Participants) | 34 | 30 | 31 | 46 | 33 | 30
Degrees Celcius | 49.9 (1.6) | 50.3 (1.7) | 50.1 (1.3) | 50.1 (1.9) | 49.8 (2.9) | 49.2 (3.5)

4. Primary Outcome: Cold Pain Tolerance - Baseline: Maximum Temperature (Cold) That Could be Tolerated by Participants
Description: Changes in response to cold stimulation stated as tolerance to cold. Responses are measured with a quantitative sensory testing (QST) device. Measurements were taken before the course of a 4 week acupuncture treatment schedule.
Time Frame: Start of Week 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees Celcius
Arm/Group | Healthy - True Acupuncture | Healthy - Sham Acupuncture | Healthy - No Treatment | Pain - True Acupuncture | Pain - Sham Acupuncture | Pain - No Treatment
Number analyzed (Participants) | 34 | 30 | 31 | 46 | 33 | 30
Degrees Celcius | 1.2 (3) | 0.5 (1) | 2.1 (5) | 2.5 (5.5) | 2.8 (6.1) | 1.1 (3.5)

5. Primary Outcome: Cold Pain Tolerance - Visit 2 or 4: Maximum Temperature (Cold) That Could be Tolerated by Participants
Description: Changes in response to cold stimulation stated as tolerance to cold. Responses are measured with a quantitative sensory testing (QST) device. Measurements were taken during the course of a 4 week acupuncture treatment schedule. Those in the no treatment groups were attending their 2nd visit, which occured on the same timeline as if they were attending the 4th visit as a treatment group subject.
Time Frame: End of Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees Celcius
Arm/Group | Healthy - True Acupuncture | Healthy - Sham Acupuncture | Healthy - No Treatment | Pain - True Acupuncture | Pain - Sham Acupuncture | Pain - No Treatment
Number analyzed (Participants) | 34 | 30 | 31 | 46 | 33 | 30
Degrees Celcius | 1.7 (4.1) | 0.3 (1.3) | 1.9 (3.9) | 2.2 (5.6) | 2.8 (5.8) | 2.4 (6.1)

6. Primary Outcome: Cold Pain Tolerance - Visit 3 or 7: Maximum Temperature (Cold) That Could be Tolerated by Participants
Description: Changes in response to cold stimulation stated as tolerance to cold. Responses are measured with a quantitative sensory testing (QST) device. Measurements were taken after the course of a 4 week acupuncture treatment schedule. Those in the no treatment groups were attending their 3rd visit, which occured on the same timeline as if they were attending the 7th visit as a treatment group subject.
Time Frame: End of Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees Celcius
Arm/Group | Healthy - True Acupuncture | Healthy - Sham Acupuncture | Healthy - No Treatment | Pain - True Acupuncture | Pain - Sham Acupuncture | Pain - No Treatment
Number analyzed (Participants) | 34 | 30 | 31 | 46 | 33 | 31
Degrees Celcius | 1.8 (4.2) | 0.1 (0.3) | 2 (4.5) | 3.7 (7.4) | 3.3 (7.1) | 1.9 (5.7)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the 4 week period that a subject was participating in the study from enrollment to completion/termination of study activities.
Arm/Group | Healthy - True Acupuncture | Healthy - Sham Acupuncture | Healthy - No Treatment | Pain - True Acupuncture | Pain - Sham Acupuncture | Pain - No Treatment
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/34 | 0/56 | 0/42 | 0/38
Other Adverse Events (participants affected / at risk) | 1/39 | 0/39 | 0/34 | 0/56 | 0/42 | 0/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy - True Acupuncture (N=39) | Healthy - Sham Acupuncture (N=39) | Healthy - No Treatment (N=34) | Pain - True Acupuncture (N=56) | Pain - Sham Acupuncture (N=42) | Pain - No Treatment (N=38)
Feeling of heaviness and muscle spasm at site of acupuncture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No